CLINICAL TRIAL: NCT05745818
Title: Colchicine for Reduction of Periprocedural Myocardial Injury in Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Tarik Mahmoud Abdellah, Dr, Sohag University
Other Study IDs: Colchicine study
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Periprocedural Myocardial Infarction; Periprocedural Myocardial Injury
Keywords: Colchicine - PCI - PPMI
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- colchicine group
  Interventions: Drug: Colchicine Pill
- control group

INTERVENTIONS:
Drug: Colchicine Pill — oral pills
  Groups: colchicine group

SUMMARY:
Study of role of colchicine in reducing periprocedural myocardial injury in patients prepared for elective PCI and its role in reduction of MACEs.

DETAILED DESCRIPTION:
Prospective open-label randomized cohort study including two groups of patients admitted and prepared for elective PCI at cardiology unit, IMD, Sohag University Hospital, these two groups are:

1. group of patients received oral tablet colchicine 6-24 hours before PCI loading dose 1 mg followed by 500 mcg after one hour.

   N.B. usual side effects of colchicine gastrointestinal disorders rarely, myalgia and weakness. Treatment of side effects symptomatic treatment ( antiemetic, etc.)
2. control group of patients. Number of patients according to sample size equation.

Sample size equation is used to calculate the minimum size of the required sample:

n = (z)2 p (1- p) / d2

* Number of patients according to sample size equation about 300 patients 150 patient in each group of study.
* Estimated study duration 2 years.
* N.B. Randomization method: first patient prepared to PCI will be included in colchicine group second patient will be included in control group and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Elective PCI in ACS patients with cardiac troponin peaked and stabilized and CCS patients .
2. PP Myocardial Injury (Any increase in post-PCI troponin if pre-PCI troponin is negative or rise in post-PCI troponin above baseline pre-PCI troponin when it is peaked and stabilized).
3. PPMI (rise in post-PCI troponin plus new evidence of ischemia).

Exclusion Criteria:

1. Patients with active infections.
2. Patients taking anti-inflammatory medications.
3. Patients presented with ACS( still rising troponin).
4. Severe renal impairment ( creatinine clearance < 45 ml/min ).
5. Primary PCI, rescue PCI, pharmacoinvasive therapy.
6. Connective tissue diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: IHD patients in IMD sohag university hospital prepared for elective PCI
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
MACEs | one month
  Major Adverse Cardiac Events

IPD SHARING:
Plan to Share IPD: Undecided